CLINICAL TRIAL: NCT02969499
Title: Electroconvulsive Therapy for Behavioural and Psychological Symptoms of Dementia: A Prospective, Open-Label, Observational Study
Brief Title: Safety and Efficacy of Electroconvulsive Therapy (ECT) for Behavioural and Psychological Symptoms of Dementia (BPSD)
Acronym: ECTBPSD
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Ontario Shores Centre for Mental Health Sciences (Other)
Responsible Party: Principal Investigator, Peter Y Chan, Clinical Professor, University of British Columbia
Other Study IDs: H15-02351
Record Dates: First submitted 2016-11-01; First posted 2016-11-21 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Dementia
Keywords: Electroconvulsive Therapy; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, open-label, observational study of the efficacy and safety of ECT for BPSD. There is no control or comparison group. Subjects will be compared on outcome measures pre- and post-ECT (and/or with a repeated measures design). Target sample size is 30 subjects over three years

DETAILED DESCRIPTION:
The study population are patients whom have a diagnosis of dementia and has behavioural and psychiatric symptoms of dementia (BPSD). In this study, the participants will have already been treated with antipsychotic medications as per usual practice but still do not have adequate symptoms control. One of the options in current clinical practice is to consider Electroconvulsive therapy (ECT) for treatment-resistant BPSD, particularly in those with psychosis and/or substantial aggression. Therefore, the study involves offering ECT to these individuals and measuring the patient's clinical status and severity of symptoms before and after ECT treatments by using standardized rating scales. Further, background information about the patient will be collected, such as their age and medical conditions.

ECT for BPSD has been done previously as reported in the medical literature. It has shown significant benefit for individuals when medication does not provide enough symptomatic relief. This research project is part of a larger multi-site study done in conjunction with Ontario Shores academic research group in Ontario, Canada. Active recruitment began in Ontario since October 2012, but our University of British Columbia (UBC) site is hoping to recruit further subjects to the total of 30 participants between the two sites.

ELIGIBILITY:
Inclusion Criteria:

* Severe BPSD: BPSD of sufficient severity that the safety of the patient or others precludes the possibility of discharge to any non-hospital environment.
* Failed "standard of care for BPSD":

  * Non-pharmacological treatments (see Clinical Practice Guideline) are of insufficient benefit to allow discharge to any non-hospital environment, and
  * Pharmacological treatments are of insufficient benefit to allow discharge to any non-hospital environment. Pharmacological treatments must consist of the following prescribed specifically for BPSD:

    * at least three atypical antipsychotic agents each for at least 4 weeks
    * at least one of the following for at least four weeks: an antidepressant, a cholinesterase inhibitor, and/or and N-methyl-D-aspartate (NMDA) receptor antagonist (i.e. memantine).
* Provided informed (substitute) consent to their attending psychiatrist for off-label treatment of BPSD with ECT as per the Health Care (Consent) and Care Facility (Admission) Act, and institutional policies and procedures.
* Been medically-cleared for ECT by Anaesthesia as per the usual pre-ECT work-up for patients admitted to the Geriatric Psychiatry Units.

Exclusion Criteria:

* Patients that are medically unfit to undergo ECT as per consultation with an anesthetist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dementia as defined by DSM-IV-TR criteria
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-11; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chan Peter, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Mount Saint Joseph's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital - Willow Pavilion, Vancouver, British Columbia
  - Ontario Shores, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: No
Data will be collected and analyzed collectively and there is no plan of making the individual data available

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: Participants recruited require a diagnosis of dementia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria (APA, 2000) and were referred to ECT for treatment of agitation and/or aggression. They have failed non-pharmacological treatments and failed at least 2 psychotropic medications at adequate dose and duration or stopped due to adverse effects. They have to be cleared by an anesthetist as being medically stable to receive ECT. Patients are excluded from the study if their temporary substitute decision make did not consent to participation in this study or they are medically unstable to receive ECT as determined by an anesthetist.
Period: Overall Study
Arm/Group | Study Participants
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 74 [66.2 to 81.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 22
  Asian | 1
  Sri Lankan | 1
  Unknown / No information | 9
Educational attainment [Count of Participants; unit: Participants]
  Below Highschool | 3
  Highschool | 11
  College | 1
  University and above | 6
  Unknown | 12
Residential setting (i.e. community vs. institutional) [Count of Participants; unit: Participants]
  Community | 2
  Instiutional | 31
Dementia type(s) [Count of Participants; unit: Participants]
  Alzheimer's | 14
  Vascular | 4
  Frontotemporal | 5
  Parkinson's | 1
  Mixed Alzheimer and Vascular | 3
  Mixed | 3
  Others | 2
  Lewy Body | 1
Dementia severity (FAST scale described below) [Mean (Standard Deviation); unit: scores on scale] — The FAST scale is a functional scale designed to evaluate patients at the more moderate-severe stages of dementia when the Mini Mental State Exam (MMSE) no longer can reflect changes in a meaningful clinical way.
  The FAST scale has seven stages:
  1. which is normal adult
  2. which is normal older adult
  3. which is early dementia
  4. which is mild dementia
  5. which is moderate dementia
  6. which is moderately severe dementia
  7. which is severe dementia
  scores on scale | 6.5 (0.54)
Previous ECT [Count of Participants; unit: Participants]
  Yes | 3
  No | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuropsychiatric Inventory (NPI)
Description: The NPI is a condition-specific measure designed to assess neuropsychiatric disturbances in people with Alzheimer Disease (AD), as well as other related dementing disorders. It assesses 12 behavioral disturbances, namely delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, aberrant motor activity, night-time behavior disturbances, and appetite / eating abnormalities. The NPI assesses not only the presence, but also the frequency and severity of each behavior. The frequency is scored from 0 (never) to 4 (very frequently). The Severity is scored from 0 (none) to 3 (marked).
  The domain score is obtained by multiplying the frequency and severity scores. The total NPI score is the sum total of all of the individual domain scores (0-144).
  NPI scores 7 days pre-ECT will be compared with NPI scores 7 days after completion of ECT course.
Time Frame: NPI measured 7 days pre-ECT and then 7 days after completing ECT course
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 33
units on a scale | -32.79 (24.72)

2. Secondary Outcome: Change in Pittsburgh Agitation Scale (PAS)
Description: The PAS assesses agitation for individuals with dementia. The scale focuses on four behaviour groups: aberrant vocalizations, motor agitation, aggressiveness and resisting care.
  Each behaviour group is measured on an intensity scale ranging from 0 (not present) -4 (extremely loud screaming or yelling, highly disruptive, unable to redirect).
  The score in each behaviour group is combined for the total PAS score of maximum 16 and minimum 0.
  PAS scores 7 days pre-ECT will be compared with scores during the ECT course and at the outlined time intervals after ECT course completion
Time Frame: For the reported value here, PAS measured 7 days pre-ECT is compared with 8 weeks after ECT course
Population: Some participants unfortunately did not have did available for analysis due to data not collected by research team staff
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 27
units on a scale | -4.83 (1.14)

3. Secondary Outcome: Change in Cornell Depression Scale (CDS) Before ECT, During Treatment Course and After Treatment Completion
Description: The Cornell Scale for Depression in Dementia (CSDD) was specifically developed to assess signs and symptoms of major depression in patients with dementia.
  Each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). The item scores are added to produce the total score. (maximum 38 and minimum 0) CDS scores 7 days pre-ECT will be compared with scores during the ECT course and 2 weeks after ECT course completion
Time Frame: For outcome report here: CDS measured 7 days pre-ECT is compared to 2 weeks after ECT course completion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 31
units on a scale | -6.26 (0.95)

4. Secondary Outcome: Change in Cornell-Brown Quality of Life Scale (CBS)
Description: The Cornell-Brown Quality of Life Scale measures quality of life in patients with dementia. It measures 19 items with score range of -2 to +2. Total score of -38 to +38 will be produced. This will be measured 7 days pre- vs. post-ECT (day 7)
Time Frame: For result reported here, CBS measured 7 days pre-ECT is compared to 7 days post ECT course completion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 31
units on a scale | 6.26 (0.95)

5. Secondary Outcome: Change in Functional Assessment Staging of Alzheimer's Disease (FAST)
Description: The FAST scale is a functional scale designed to evaluate patients at the more moderate-severe stages of dementia when the MMSE no longer can reflect changes in a meaningful clinical way.
  The FAST scale has seven stages:
  1. which is normal adult
  2. which is normal older adult
  3. which is early dementia
  4. which is mild dementia
  5. which is moderate dementia
  6. which is moderately severe dementia
  7. which is severe dementia
  FAST score 7 days pre-ECT will be compared with score during ECT course and up to 8 weeks after course completion as outlined
Time Frame: For outcome reported here, FAST measured 7 days pre-ECT is compared to 8 weeks after completion of ECT course
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 33
units on a scale | 0.12 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse effects are collected by using the Columbia ECT subjective side effect schedule. This 32 item scale will be administered at baseline (7 days pre-ECT) and in the afternoon following the 1st, 4th and 8th treatments and in the week following the course of ECT (post-treatment day 7).
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 1/33
Other Adverse Events (participants affected / at risk) | 5/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=33)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient passed away 2 days after their last ECT due to pneumonia but it was felt that was unlikely to be directly related to ECT treatment as the patient was frail
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=33)
Delirium (Renal and urinary disorders) | 2 (2) — Two participants had ECT held temporarily due to increased confusion when they developed a urinary tract infection. The delirium in each was not deemed to be related to ECT.
Agitation (Nervous system disorders) | 2 (2) — Two participants manifested agitation/restlessness after ECT, and it was not clear if this represented an exacerbation of their (Neuro-Psychiatric Symptoms) NPS or if there was concurrent transient post-ECT delirium.
Hypotension/Bradycardia (Cardiac disorders) | 1 (1) — One participant had a transient bout of hypotension and bradycardia after an ECT treatment

LIMITATIONS AND CAVEATS:
Retrospective design, medication use not controlled for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT02969499/Prot_SAP_000.pdf